CLINICAL TRIAL: NCT04683367
Title: 15-year Follow-up of Laparoscopically Diagnosed Occult Inguinal and Ventral Hernias
Brief Title: Follow-up of Symptomless Inguinal and Ventral Hernias
Acronym: hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Hannu Paajanen, Professor of Surgery, Kuopio University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 139/2020
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Hernia, Inguinal; Hernia, Ventral; Laparoscopy
Keywords: inguinal hernia; ventral hernia; laparoscopic diagnosis
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral | interventions — Laparoscopy; Herniorrhaphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- clinical hernia (Experimental): developing clinical hernia
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — laparoscopic repair of hernia
  Other Names: hernioplasty

SUMMARY:
The orifices of all inguinal and ventral (including Spigelian) hernias were carefully recorded at the beginning of laparoscopy (n=201) of other reason (cholecystectomy, fundoplication) in 2003-5. The patients with occult hernias (n=43) were followed-up 15 years to find out what percentage of hernias would become symptomatic.

DETAILED DESCRIPTION:
This was a prospective laparoscopic study of 201 consecutive adult patients operated in 2003-5. There were 133 females and 68 males with a mean age 53 ± 14 years. The index laparoscopic operation included 104 cholecystectomies, 55 fundoplications, 36 diagnostic, 5 appendectomies and one insertion of peritoneal catheter. A careful clinical examination of the groin and ventral region was performed on everybody and all patients with clinical hernias were excluded. Laparoscopic exploration of the inguinal region was considered safe and did not greatly increase the operative time. All patients were informed that hernial orifices would be explored during laparoscopy, and a written consent was asked prior to surgery. Permission to repair large hernias (> 1 cm) was also obtained before laparoscopy.

The patients were followed-up 15 years to find out, what percentage of occult, symptomless inguinal and ventral hernias were later operated because of harmfull symptoms.

ELIGIBILITY:
Inclusion Criteria:

* occult inguinal or ventral hernia diagnosed in laparoscopic surgery

Exclusion Criteria:

* clinically diagnosed inguinal or ventral hernia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
number of operated hernia | 15 years
  occult hernia operated because of symptoms

SECONDARY OUTCOMES:
number of symptomatic hernia | 15 years
  incipient, asymptomatic hernia becomes symptomatic during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hannu EK Paajanen, MD, PhD, Principal Investigator — department of Surgery, Kuopio Univ Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland